CLINICAL TRIAL: NCT00928239
Title: Laparoscopic Sacropexy: Randomized Clinical Trial to Compare Two Different Attachment Sites of the Dorsal Mesh at the Vaginal Insertion(MeshPlace)
Brief Title: Laparoscopic Sacropexy: Comparison of Mesh Attachment
Acronym: MeshPlace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Dimitri Sarlos, Department of Gynecology and Obstetrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSA-MeshPlace
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Vaginal Vault Prolapse
Keywords: vaginal vault prolapse; laparoscopic sacropexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Arm1: Laparoscopic repair of vaginal vault prolapse. Laparoscopic sacropexy procedure as described in previous publication(Sarlos D, Brandner S, Kots L, Gygax N, Schaer G. Laparoscopic sacrocolpopexy for uterine and post-hysterectomy prolapse: anatomical results, quality of life and perioperative outcome-a prospective study with 101 cases. Int Urogynecol JPelvic Floor Dysfunct. 2008 Oct;19(10):1415-22. Epub 2008 Jun 7. PubMed PMID: 18536861) with attachment to the caudal part of the vagina and the apex.
  Interventions: Procedure: laparoscopic sacropexy with mid vaginal attachment
- 2 (Active Comparator): Arm 2: Laparoscopic repair of vaginal vault prolapse. Laparoscopic sacropexy procedure as described in previous publication(Sarlos D, Brandner S, Kots L, Gygax N, Schaer G. Laparoscopic sacrocolpopexy for uterine and post-hysterectomy prolapse: anatomical results, quality of life and perioperative outcome-a prospective study with 101 cases. Int Urogynecol JPelvic Floor Dysfunct. 2008 Oct;19(10):1415-22. Epub 2008 Jun 7. PubMed PMID: 18536861) with attachment of the dorsal mesh at distal end of vagina at dorsal vaginal wall
  Interventions: Procedure: laparoscopic sacropexy with caudal vaginal attachment

INTERVENTIONS:
Procedure: laparoscopic sacropexy with mid vaginal attachment — * supracervical hysterectomy for uterine prolapse
  * exposure of the anterior longitudinal ligament of sacrum and recto-vaginal septum posterior
  * dissection up to ventrolateral part of the levator ani muscle
  * Anterior dissection of vesico-vaginal fascia up to the lower third of the vagina below the trigonum of bladder
  * Two separate meshes, Gynemesh® (Johnson&Johnson) a polypropylene mesh, for anterior and posterior compartment
  * suturing of posterior mesh caudally to levator ani muscle and proximally 4cm from the apex of the vagina or cervical stump
  * placement of anterior mesh underneath bladder and attachment to caudal part of the vagina and the apex
  * suturing together anterior and posterior mesh are sutured together at level of vaginal apex and attachment to longitudinal sacral ligament at level of S2
  Other Names: laparoscopic sacrocolpopexy
  Arms: 1
Procedure: laparoscopic sacropexy with caudal vaginal attachment — * supracervical hysterectomy for uterine prolapse
  * exposure of the anterior longitudinal ligament of sacrum and recto-vaginal septum posterior
  * dissection up to ventrolateral part of the levator ani muscle
  * Anterior dissection of vesico-vaginal fascia up to the lower third of the vagina below the trigonum of bladder
  * Two separate meshes, Gynemesh® (Johnson&Johnson) a polypropylene mesh, for anterior and posterior compartment
  * suturing of posterior mesh caudally to the levator ani muscle and proximally at caudal part of the vagina or cervical stump
  * placement of anterior mesh underneath bladder and attachment to caudal part of the vagina and the apex
  * suturing together anterior and posterior mesh are sutured together at level of vaginal apex and attachment to longitudinal sacral ligament at level of S2
  Other Names: laparoscopic sacrocolpopexy
  Arms: 2

SUMMARY:
The purpose of this study is to compare postoperative complications and outcome two different attachment sites of the dorsal mesh support in laparoscopic sacropexy.

DETAILED DESCRIPTION:
Laparoscopic sacropexy has become a well established treatment option for vaginal vault prolapse with excellent outcome and low rates of recurrence. Compared to the similar vaginal sacropexy procedure a significant rate of postoperative constipation is reported. As the surgical technique is very similar for both procedures it could be possible that the exposure of the lower vaginal wall and placement and of the dorsal mesh and closer proximity to the colon in laparoscopic sacropexy might cause this. In this randomized controlled clinical trial we compare two different attachment sites for the dorsal mesh during laparoscopic sacropexy. One group is randomized for attachment in the middle of the dorsal wall of the vaginal stump and for the other group preparation and attachment for the dorsal mesh is performed deeper in the lower pelvis for an attachment at the distal part of the dorsal vaginal wall.

Peri-operative data, intra- and postoperative complications and results of short-term (constipation) and long-term( recurrences rate) outcome are recorded.

ELIGIBILITY:
Inclusion Criteria:

* vaginal vault prolapse
* recurrence of vaginal vault prolapse
* signed consent

Exclusion Criteria:

* rectocele
* BMI>40

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Constipation | 6 to 8 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Sarlos, MD, Study Chair — Kantonsspital Aarau, Department of Gynecology and Obstetrics
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland